CLINICAL TRIAL: NCT02817386
Title: microRNA and Delirium After Hip and Knee Fracture
Brief Title: Study of Postoperative Delirium in Elderly People After Orthopedic Surgery
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Mian Peng,MD, vice professor, Zhongnan Hospital
Other Study IDs: 2015002
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Postoperative Delirium
Keywords: postoperative delirium; microRNA
MeSH Terms: conditions — Emergence Delirium | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- POD and Non-POD;: Trained clinical research assistants interviewed the patients on the first and second day post surgery. The assessment of post deliriu (POD) was performed once per day between 8:00 AM to 10:00 AM. Patient notes were not reviewed for episodes of delirium which could occur outside the time of assessment. The clinical research assistants who performed the delirium assessments in this study had good training and went through quality control procedures. We used state-of-the-art delirium detection methods, which tend to report a higher incidence of delirium. The interview included the Confusion Assessment Method (CAM) and Memorial Delirium Assessment Scale (MDAS).
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — Trained clinical research assistants interviewed the patients on the first and second day post surgery. The interview included the Confusion Assessment Method (CAM) and MDAS. CAM is a diagnostic algorithm used to determine the presence or absence of delirium.

SUMMARY:
The purpose of this study is to investigate the possible relationship of microRNA and postoperative delirium.

DETAILED DESCRIPTION:
Postoperative delirium is one of the most common postoperative complications in elderly patients.It has been shown that postoperative delirium has independent adverse effects on short and long-term mortality and morbidity, including poor functional recovery, postoperative cognitive dysfunction, deterioration in quality of life, and increased costs. However, at the present time, postoperative delirium is a clinical phenomenon, and its neuropathogenesis remains unknown. This gap in knowledge has become a barrier that limits further studies, including the development of potential interventions for postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years old or older
2. candidates for spinal anesthesia
3. Non language communication barriers

Exclusion Criteria:

1. past medical history of neurological and psychiatric diseases including AD, other forms of dementia, stroke, or psychosis;
2. severe visual or hearing impairment;
3. unwillingness to comply with the protocol or procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A total of 60 adults who were scheduled to have elective total hip or knee replacement surgery at the Zhongnan Hospital were asked to participate in this study.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-03; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The level of microRNA in cerebrospinal fluid and serum | through study completion, an average of 1 year
  All of the participants had spinal anesthesia for the scheduled surgery. Two milliliter of CSF was collected from a spinal needle by anesthesiologists during the spinal anesthesia before the administration of the local anesthetic. Blood samples were collected from patients prior to spinal anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Mian Peng, MD, Study Director — Zhongnan Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xie Z, Swain CA, Ward SA, Zheng H, Dong Y, Sunder N, Burke DW, Escobar D, Zhang Y, Marcantonio ER. Preoperative cerebrospinal fluid beta-Amyloid/Tau ratio and postoperative delirium. Ann Clin Transl Neurol. 2014 May 1;1(5):319-328. doi: 10.1002/acn3.58. PMID 24860840
- [Derived] Dong R, Sun L, Lu Y, Yang X, Peng M, Zhang Z. NeurimmiRs and Postoperative Delirium in Elderly Patients Undergoing Total Hip/Knee Replacement: A Pilot Study. Front Aging Neurosci. 2017 Jun 23;9:200. doi: 10.3389/fnagi.2017.00200. eCollection 2017. PMID 28690539